CLINICAL TRIAL: NCT06035523
Title: A Single Arm Pilot Study Evaluating Wound Closure With a Unique Staged Application of Endoform™ and Symphony™ in the Treatment of Non-Healing Diabetic Foot Ulcers
Brief Title: Clinical Study Evaluating Wound Closure With Endoform™ and Symphony™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aroa Biosurgery Limited (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AROA 002
Record Dates: First submitted 2023-08-23; First posted 2023-09-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Wound Healing; Diabetic Foot; Chronic Foot Ulcer; Foot Ulcer
Keywords: Extracellular matrix; Regenerative medicine; Leg ulcer; Diabetes complications; Diabetic Angiopathies; Diabetes Mellitus
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Leg Ulcer; Diabetes Complications; Diabetic Angiopathies; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects with a Wagner Grade 1 or 2 diabetic foot ulcer (Other): Arm receives application of Endoform™ Antibacterial, Endoform™ Natural and Symphony™ and appropriate Off - loading
  Interventions: Device: Endoform™ Antibacterial; Device: Endoform™ Natural; Device: Symphony™

INTERVENTIONS:
Device: Endoform™ Antibacterial — Application of Endoform™ Antibacterial
Device: Endoform™ Natural — Application of Endoform™ Natural
Device: Symphony™ — Application of Symphony™

SUMMARY:
Study will evaluate the performance and safety of Endoform™ Natural and Endoform™ Antimicrobial in conjunction with Symphony™ in the treatment of chronic non-healing diabetic foot ulcers after 12 weeks of treatment.

DETAILED DESCRIPTION:
About 50 subjects will take part in this study. The purpose of this study is to evaluate the performance and safety of Endoform™ Natural and Endoform™ Antimicrobial in conjunction with Symphony™ (together, the 'Products') in the treatment of acute or chronic non-healing wounds, including diabetic foot ulcers Wagner Grade 1 or 2, after 12 weeks of treatment.

Following initial enrollment, eligible subjects will then undergo

* a treatment phase involving weekly treatment and evaluations for up to 12 weeks,
* subjects that heal will enter a follow-up period that includes 1 visit (Healing Confirmation Visit), 2 weeks from initial healing.
* If the subject does not heal, they will exit at Week 13, End of Study visit.

All subjects will require accepted routine procedures as part of standard of care (SOC): offloading of the DFU (removeable cast boot or total contact casting [TCC] if the subject's foot is too large for a removeable cast boot), appropriate sharp debridement, and infection management. In addition, each subject will receive a wound care covering comprising of either Endoform™ Antimicrobial, Endoform™ Natural or Symphony™ followed by a silicone non-adherent dressing (MepitelTM or equivalent), a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll, compressive wrap and Coban (Threeflex 3-layer or equivalent).

ELIGIBILITY:
Inclusion Criteria:

* 1. At least 18 years old, inclusive.
* 2. Presence of a DFU, Wagner Grade 1 or 2 (see Appendix D for definitions), extending through the dermis provided it is below the medial aspect of the malleolus.
* 3. The index ulcer (ulcer to be evaluated in the study) will be the largest ulcer if two or more DFUs are present with the same Wagner grade and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
* 4. Index ulcer has been present for greater than 4 weeks prior to SV1 and less than 1 year, as of the date the subject consents for study.
* 5. Index ulcer is a minimum of 1.0 cm2 and a maximum of 25 cm2 at SV1 and TV1.
* 6. Within 3 months of SV1, adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) between 0.7 and 1.3 using the affected study extremity. As an alternative, arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of > 0.6 is acceptable.
* 7. The target ulcer has been offloaded for at least 14 days, prior to SV1.
* 8. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
* 9. Subject understands and is willing to participate in the clinical study and can comply with weekly visits.
* 10. Subjects must have read and signed the IRB approved ICF before screening procedures are performed.

Exclusion Criteria:

* 1. Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
* 2. Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
* 3. Index ulcer is overtly infected (i.e., purulent drainage).
* 4. Subjects with a history of more than two weeks of treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study.
* 5. Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1.
* 6. History of radiation at the ulcer site (regardless of time since last radiation treatment).
* 7. Index ulcer has been previously treated or will need to be treated with any prohibited therapies.
* 8. Subjects with a previous diagnosis of HIV or Hepatitis C.
* 9. Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
* 10. Osteomyelitis or bone infection of the affected foot as verified by xray within 30 days prior to the first screening visit. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).
* 11. Subject is pregnant or breast-feeding.
* 12. Presence of diabetes with poor metabolic control as documented with an HbA1c >12.0 within last 90 days.
* 13. Subjects with end stage renal disease as evidenced by a serum creatinine ≥3.0 mg/dL within 6 months of enrollment
* 14. Presence of acute Charcot Neuroarthropathy to the affected limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
Percentage of index ulcers (the ulcers being treated in the study) healed at 12 weeks | 12 weeks
  Percentage of index ulcer defined as 100% re-epithelialization within 12 weeks

SECONDARY OUTCOMES:
Time to heal within 12 weeks | 12 weeks
  Time to heal of index ulcer defined as 100% re-epithelialization within 12 weeks
Percentage area reduction at 12 weeks | 12 weeks
  Area reduction percentage of ulcers at 12 weeks
Changes in wound quality of life (per W-QoL) | 12 weeks
  Changes in wound quality of life (W-QoL), using the W-QoL short questionnaire administered on Study Visit 1 (as a baseline) and after 12 weeks of treatment (End of Study Visit). Each item is scored on a 5-point Likert scale from 0 (not at all) to 4 (very much).
Change in subjects reported pain levels (NPRS) | 12 weeks
  Change in subject-reported pain levels using the 0-10 Numeric Pain Rating Scale at baseline (Study Visit 1) and after 12 weeks of treatment EOS visit (End of Study Visit).On the numerical pain scale, the number 0 represents "no pain" and the number 10 represents "the worst possible pain".

OTHER OUTCOMES:
Product wastage | 12 weeks
  For each product, the size actually used will be the basis to calculate the area of the product.
  Based on the investigator's notes, wound area at time of application will be calculated as a rectangle (length x width) reduced to an ellipsoid.
  Wastage = ((area of product - area of wound)/area of product)*100
Cost to closure | 12 weeks
  Calculation of cost of treatment, including number of device applications for each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, DPM, MD PhD, Study Chair — Keck School of Medicine
Locations (4):
- United States (4):
  - South Florida Lower Extremity Center, Hollywood, Florida
  - Advanced Pharma Cr, LLC, Miami, Florida
  - Foot and Ankle Specialists of the Mid-Atlantic, Salem, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No